CLINICAL TRIAL: NCT03035058
Title: A Randomized, Global, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate the Efficacy and Safety of Vedolizumab IV for the Treatment of Primary Sclerosing Cholangitis, With Underlying Inflammatory Bowel Disease
Brief Title: Efficacy and Safety of Vedolizumab Intravenous (IV) in the Treatment of Primary Sclerosing Cholangitis in Subjects With Underlying Inflammatory Bowel Disease
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MLN0002-3023; 2014-003942-28 (EudraCT Number); U1111-1161-4900 (Registry Identifier: WHO); 16/LO/0288 (Registry Identifier: NRES); NL56650.056.16 (Registry Identifier: CCMO); 191059 (Registry Identifier: HC-CTD)
Record Dates: First submitted 2017-01-25; First posted 2017-01-27 (Estimated); Last update posted 2017-03-08 (Actual); Status verified 2017-03

CONDITIONS: Primary Sclerosing Cholangitis; Inflammatory Bowel Disease
Keywords: Drug therapy
MeSH Terms: conditions — Cholangitis, Sclerosing; Inflammatory Bowel Diseases | interventions — vedolizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Vedolizumab IV 300 mg Q4W (Experimental): Vedolizumab 300 mg, intravenous (IV), once at Day 1 and Week 2; followed by vedolizumab 300 mg, IV, once every 4 weeks (Q4W) starting from Week 6 to Week 102.
  Interventions: Drug: Vedolizumab
- Vedolizumab IV 300 mg Q8W + Placebo (Experimental): Vedolizumab 300 mg, IV, once at Day 1 and Week 2; followed by vedolizumab 300 mg, IV, once every 8 weeks (Q8W) starting from Week 6 to Week 102 (and placebo, IV, Q8W starting from Week 10 to Week 98.
  Interventions: Drug: Vedolizumab; Drug: Placebo
- Placebo (Placebo Comparator): Vedolizumab placebo-matching, IV, at Day 1 and Week 2; followed by Vedolizumab placebo-matching, IV, Q4W starting from Week 6 to Week 102.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vedolizumab — Vedolizumab intravenous infusion
  Other Names: MLN0002; ENTYVIO; KYNTELES
  Arms: Vedolizumab IV 300 mg Q4W; Vedolizumab IV 300 mg Q8W + Placebo
Drug: Placebo — Placebo
  Arms: Placebo; Vedolizumab IV 300 mg Q8W + Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of vedolizumab intravenous (IV) in non-end-stage primary sclerosing cholangitis (PSC) participants with underlying inflammatory bowel disease (IBD).

DETAILED DESCRIPTION:
The drug being tested in this study is called vedolizumab. Vedolizumab is being tested to treat people who have non-end-stage primary sclerosing cholangitis (PSC) with underlying inflammatory bowel disease (IBD). This study will look at changes in fibrosis staging in people who take vedolizumab.

The study will enroll approximately 258 patients. Participants will be randomly assigned (by chance, like flipping a coin) to one of the three treatment groups in ratio 1:1:1-which will remain undisclosed to the patient and study doctor during the study (unless there is an urgent medical need):

* Vedolizumab 300 mg once every 4 weeks (Q4W)
* Vedolizumab 300 mg once every 8 weeks (Q8W)
* Placebo (dummy inactive pill) - this is a tablet that looks like the study drug but has no active ingredient

All participants will be administered vedolizumab or placebo via intravenous infusion

This multi-center trial will be conducted worldwide. The overall time to participate in this study is up to 124 weeks. Participants will make multiple visits to the clinic and will be contacted by telephone 6 months after last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Has chronic cholestatic liver disease, of at least 6 months duration, with a subsequent diagnosis of primary sclerosing cholangitis (PSC), based on cholangiographic findings of intrahepatic and/or extrahepatic bile duct irregularities consistent with PSC.
2. Has a diagnosis of inflammatory bowel disease (IBD) (either ulcerative colitis [UC], Crohn's disease [CD], or IBD unclassified [IBDU]), established at least 3 months prior to enrollment by clinical and endoscopic evidence and corroborated by a histopathology report.
3. Has a liver stiffness transient elastography (TE) score of ≤14.3 kPa, as assessed by FibroScan.
4. Has had a colorectal cancer screen within 12 months of the Screening Visit with no signs of malignancy, dysplasia, or neoplasia.

Exclusion Criteria:

Hepatic and Gastrointestinal Exclusion Criteria

1. Has received any fibrates within 8 weeks of Screening.
2. Has high suspicion of cholangiocarcinoma, as indicated by an elevated Ca 19-9 value (>129 U/mL) at screening.
3. Has evidence of overlap syndrome with autoimmune hepatitis or primary or secondary biliary cirrhosis or autoimmune cholangitis, as judged by the investigator.
4. Has evidence of alcoholic liver disease including history of alcoholic hepatitis.
5. Has a diagnosis of small duct PSC.
6. Has a Model for End-Stage Liver Disease (MELD) score >12 at screening.
7. Has a Child-Pugh score >7 (following adjustment for PSC diagnosis) at screening.
8. Has received a liver transplant.
9. Has evidence of autoimmune immunoglobin (Ig) IgG4-associated cholangitis, as defined by elevated serum IgG4 at least 2 x ULN (at screening), or IgG4/IgG1 ratio above 0.24.
10. Has undergone prior biliary surgery (laparoscopic or open surgery). Participants who have undergone cholecystectomy without surgical complications will be allowed provided the surgery was not done within 6 weeks prior to screening.
11. Has had 2 or more interventional treatments for dominant stricture (including stent placement/replacement) within 12 months prior to the Screening Visit.
12. Has evidence of cholangitis, requiring antibiotics, within 3 months prior to the Screening Visit [short courses of antibiotics for no more than 5 days are allowed for stent placement or endoscopic retrograde cholangiopancreatography (ERCP) prophylaxis].

    Infectious Disease Exclusion Criteria
13. Has chronic hepatitis B virus (HBV) or hepatitis C virus (HCV) infection.
14. Has positive hepatitis B core antibody (anti-HBc) at screening.
15. Has evidence of an active infection during the Screening Period.
16. Has any identified congenital or acquired immunodeficiency (eg, common variable immunodeficiency, human immunodeficiency virus [HIV] infection, organ transplantation).
17. Has active or latent tuberculosis (TB), regardless of treatment history, as evidenced by any of the following:

    1. History of TB.
    2. A positive diagnostic TB test within 30 days of enrollment defined as: 1. A positive QuantiFERON test or 2 successive indeterminate QuantiFERON tests (or, a positive T-SPOT TB test [Japan only]), OR
    3. Chest X-ray within 3 months of enrollment in which active or latent pulmonary TB cannot be excluded

    General Exclusion Criteria
18. Has had previous exposure to natalizumab, efalizumab, rituximab, or any other integrin antagonist.
19. Has received any of the following for the treatment of underlying disease within 30 days of screening:

    * Nonbiologic therapies (eg, cyclosporine, tacrolimus, thalidomide) other than those specifically listed in the protocol for the treatment of IBD.
    * An approved nonbiologic therapy in an investigational protocol.
20. Has, in the judgment of the investigator, clinically significant abnormal hematological parameters of hemoglobin, hematocrit, or erythrocytes at the Screening Visit.
21. Has any history of malignancy, except for the following: (a) adequately treated nonmetastatic basal cell skin cancer; (b) squamous cell skin cancer that has been adequately treated and that has not recurred for at least 1 year prior to randomization; and (c) history of cervical carcinoma in situ that has been adequately treated and that has not recurred for at least 3 years prior to randomization. Participant with remote history of malignancy (eg, >10 years since completion of curative therapy without recurrence) will be considered based on the nature of the malignancy and the therapy received and must be discussed with the sponsor on a case-by-case basis prior to randomization.
22. Has a history of any major neurological disorders, including stroke, multiple sclerosis, brain tumor, demyelinating or neurodegenerative disease.
23. Has a positive response on the progressive multifocal leukoencephalopathy (PML) subjective symptom checklist prior to the administration of study drug.
24. Has received any of the following for the treatment of underlying disease within 30 days of screening:

    * Nonbiologic therapies (eg, cyclosporine, tacrolimus, thalidomide) other than those specifically listed in the protocol for the treatment of IBD.
    * An approved nonbiologic therapy in an investigational protocol.
25. Has had any surgical procedure requiring general anesthesia within 30 days prior to screening or is planning to undergo major surgery during the study.
26. Is required to take excluded medications.
27. Has received any live vaccinations within 30 days prior to screening.
28. Has evidence of or treatment for C. difficile infection within 60 days or other intestinal pathogen within 30 days prior to the Screening Visit or other known infectious, immunologic, or ischemic liver or intestinal disease that, in the investigator's opinion, may interfere with the study procedures or study results.
29. Has, in the judgment of the investigator, clinically significant abnormal hematological parameters of hemoglobin, hematocrit, or erythrocytes at the Screening Visit.
30. Has previous history of colectomy.
31. In the opinion of the investigator, the participant has a life expectancy or anticipated need for liver transplantation within <24 months.
32. Has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse within 1 year prior to screening.
33. For the magnetic resonance elastography (MRE) substudy, participants are excluded if they have contraindications to magnetic resonance (MR) scanning. Contraindications include ferromagnetic foreign bodies (eg, shrapnel, ferromagnetic fragments in the orbital area, certain tattoos), certain implanted medical devices (eg, aneurysm clips, cardiac pacemakers) or claustrophobia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-02; Primary Completion 2020-09 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with No Worsening in Ishak Fibrosis Staging Score from Baseline to Week 106 Visit | Baseline and Week 106
  Assessments will be performed from liver biopsies with histology assessed by 2 independent blinded central readers for Ishak fibrosis staging score. Ishak fibrosis staging scoring is as follows: 0=No fibrosis, 1=Fibrous expansion of some portal areas with or without septa, 2=Fibrous expansion of most portal areas with or without septa, 3=Fibrous expansion of most portal areas with occasional portal to portal bridging, 4=Fibrous expansion of portal areas with marked bridging (portal to portal and/or portal to central), 5=Marked bridging with occasional nodules (incomplete cirrhosis), 6=Cirrhosis, probable or definitive. A negative change from Baseline indicates improvement.

SECONDARY OUTCOMES:
Percentage of Participants with a ≥35% Reduction in Serum Alkaline Phosphatase (ALP) from Baseline to Week 106 Visit | Baseline and Week 106
  Blood will be collected and ALP will be assessed as part of the serum chemistry testing.
Change in Ishak Necroinflammatory Grading Score from Baseline to the Week 106 Visit | Baseline and Week 106
  Assessments will be performed from liver biopsies with histology assessed by 2 independent blinded central readers for Ishak fibrosis staging score. Ishak necroinflammatory grading score is based on assessments from 4 subscales: (A) Periportal or periseptal interface hepatitis (piecemeal necrosis) 5-point subscale (0=Absent to 4=Severe), (B) Confluent necrosis 7-point subscale (0=Absent to 6=Panacinar or multiacinar necrosis), (C) Focal (spotty) lytic necrosis, apoptosis and focal inflammation 5-point subscale (0=Absent to 4=More than ten foci per times 10 objective), and (D) Portal inflammation (0=Absent to 4=Marked, all portal areas). A negative change from Baseline indicates improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda